CLINICAL TRIAL: NCT01017874
Title: A Randomized Ph 3 Study Comparing First-Line Pemetrexed/Cisplatin Followed by Gefitinib With Gefitinib Alone in East Asian Never Smoker or Light Ex-Smoker Patients With Locally Advanced or Metastatic Nonsquamous NSCLC
Brief Title: A Study of Alimta/Cisplatin/Gefitinib for Asian Non-smoking Participants With Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13021; H3E-CR-S131 (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed + Cisplatin + Gefitinib (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Gefitinib
- Gefitinib (Active Comparator)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Pemetrexed — 500 milligrams per square meter (mg/m²) administered intravenously on Day 1 of each 21-day cycle, for 6 cycles.
  Other Names: Alimta; LY231514
  Arms: Pemetrexed + Cisplatin + Gefitinib
Drug: Cisplatin — 75 mg/m² administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
  Arms: Pemetrexed + Cisplatin + Gefitinib
Drug: Gefitinib — 250 milligrams (mg) administered orally once a day, every day of 21-day cycle, for maintenance in participants with non-progressive disease after cisplatin/pemetrexed chemotherapy
  Arms: Pemetrexed + Cisplatin + Gefitinib
Drug: Gefitinib — 250 milligrams (mg) administered orally once a day, every day of 21-day cycles administered as a monotherapy
  Arms: Gefitinib

SUMMARY:
The purpose of this study is to compare two different approaches to treating non-small cell lung cancer (NSCLC) in East Asian never-smoker participants. Half of the participants will receive chemotherapy (pemetrexed/cisplatin) followed by an oral anti-cancer agent (gefitinib) and the other half of the participants will receive only the oral anti-cancer agent (gefitinib).

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of NSCLC with locally advanced or metastatic disease that is of non-squamous histology.
* Participants must be "light ex-smokers" or "never-smokers".

  * "Light ex-smokers" defined as having ceased smoking for greater than or equal to 5 years and not to have exceeded 10 pack-years.
  * "Never-smokers" are defined as having smoked <100 cigarettes or equivalent during his/her lifetime.
* Participants must be of East Asian ethnicity.
* No prior systemic therapy for lung cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Presence of clinically significant (by physical exam) third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
* Any evidence of clinically active interstitial lung disease. Asymptomatic participants with chronic, stable, radiographic changes are eligible.
* Participants whose Epidermal Growth Factor Receptor (EGFR) mutation status is known prior to study entry will be excluded. Participants in which EGFR mutation testing has not been performed, or whose EGFR mutation status is unknown or inconclusive at study entry are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kowloon, Hong Kong
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liouying/Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puzih City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Thailand (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangkok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiang Mai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hat Yai

REFERENCES:
- [Derived] Yang JC, Srimuninnimit V, Ahn MJ, Lin CC, Kim SW, Tsai CM, Mok T, Orlando M, Puri T, Wang X, Park K. First-Line Pemetrexed plus Cisplatin followed by Gefitinib Maintenance Therapy versus Gefitinib Monotherapy in East Asian Never-Smoker Patients with Locally Advanced or Metastatic Nonsquamous Non-Small Cell Lung Cancer: Final Overall Survival Results from a Randomized Phase 3 Study. J Thorac Oncol. 2016 Mar;11(3):370-9. doi: 10.1016/j.jtho.2015.11.008. Epub 2015 Dec 25. PMID 26725183
- [Derived] Kang JH, Ahn MJ, Kim DW, Cho EK, Kim JH, Shin SW, Wang X, Kim JS, Orlando M, Park K. Tolerability and Outcomes of First-Line Pemetrexed-Cisplatin Followed by Gefitinib Maintenance Therapy Versus Gefitinib Monotherapy in Korean Patients with Advanced Nonsquamous Non-small Cell Lung Cancer: A Post Hoc Descriptive Subgroup Analysis of a Randomized, Phase 3 Trial. Cancer Res Treat. 2016 Apr;48(2):458-64. doi: 10.4143/crt.2015.135. Epub 2015 Oct 14. PMID 26511807
- [Derived] Yang JC, Kang JH, Mok T, Ahn MJ, Srimuninnimit V, Lin CC, Kim DW, Tsai CM, Barraclough H, Altug S, Orlando M, Park K. First-line pemetrexed plus cisplatin followed by gefitinib maintenance therapy versus gefitinib monotherapy in East Asian patients with locally advanced or metastatic non-squamous non-small cell lung cancer: a randomised, phase 3 trial. Eur J Cancer. 2014 Sep;50(13):2219-30. doi: 10.1016/j.ejca.2014.05.011. Epub 2014 Jun 18. PMID 24953333

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died or continued on study but discontinued receiving study drug were considered to be completed.
Groups:
- Pemetrexed + Cisplatin + Gefitinib: Pemetrexed: 500 milligrams per square meter (mg/m²) administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
  Cisplatin: 75 mg/m² administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
  Gefitinib: 250 milligrams (mg) administered orally once a day, every day of 21-day cycle, as maintenance therapy in participants with non-progressive disease after cisplatin/pemetrexed chemotherapy
- Gefitinib: Gefitinib: 250 mg administered orally once a day, every day of 21-day cycle, as a monotherapy
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Started | 118 | 118
Received at Least 1 Dose of Study Drug | 114 | 118
Completed | 88 | 92
Not Completed | 30 | 26
Not completed — Withdrawal by Subject | 23 | 20
Not completed — Sponsor decision | 3 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib | Total
Number analyzed (Participants) | 118 | 118 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.53 (10.730) | 59.36 (10.672) | 58.95 (10.686)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 89 | 177
  Male | 30 | 29 | 59
Race/Ethnicity, Customized [Number; unit: participant]
  Asian | 118 | 118 | 236
Region of Enrollment [Number; unit: participants]
  Hong Kong | 3 | 7 | 10
  Taiwan | 39 | 28 | 67
  Thailand | 21 | 22 | 43
  Singapore | 1 | 1 | 2
  Korea, Republic of | 54 | 60 | 114

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of randomization to the objective disease progression or death due to any cause. Response was defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. Progressive disease (PD) was defined as at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions. Participants who did not have a complete baseline disease assessment were censored at the date of randomization, regardless if PD was objectively determined or if participant died or if a participant was not known to have died or have objective PD at the data inclusion cutoff date. PFS was censored at the last complete objective progression-free disease assessment date.
Time Frame: Randomization to the first date of measured PD or death up to 37.32 months
Population: Intent-to-treat (ITT) population: All data from all randomized participants according to the treatment they were assigned. Censored participants: Pemetrexed+Cisplatin+Gefitinib=32, Gefitinib=22.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 118 | 118
months | 8.38 [6.44 to 11.14] | 9.63 [6.74 to 11.10]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin + Gefitinib vs Gefitinib; Test type: Superiority or Other; p = 0.217, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.63 to 1.13]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was the duration from randomization to the date of death from any cause. For participants who were not known to have died as of the data-inclusion cut-off date for a particular analysis, OS was censored at the date of last contact prior to the data inclusion cutoff date (contacts considered in the determination of last contact date included adverse event date, lesion assessment date, visit date, and last known alive date).
Time Frame: Randomization up to date of death from any cause up to 57.13 months
Population: ITT population: All data from all randomized participants according to the treatment they were assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 118 | 118
months | 26.87 [20.76 to 35.12] | 27.86 [21.26 to 31.36]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin + Gefitinib vs Gefitinib; Test type: Superiority or Other; p = 0.788, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.68 to 1.31]

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Tumor Response Rate (TRR)]
Description: TRR was defined as the percentage of randomized participants having a best overall study response of CR or PR using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all target lesions; PR was defined as at least a 30% decrease in sum of longest diameter (LD) of target lesions taking as reference the baseline sum LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions and the appearance of no new lesions.
Time Frame: Randomization up to 37.52 months
Population: Intent-to-treat (ITT) population: All data from all randomized participants according to the treatment they were assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 118 | 118
percentage of participants | 41.5 [32.5 to 51.0] | 47.5 [38.2 to 56.9]

4. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD) [Disease Control Rate (DCR)]
Description: DCR was defined as the percentage of randomized participants with overall response of CR, PR or SD using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all tumor lesions; PR was defined as at least a 30% decrease in sum of longest diameter (LD) of target lesions taking as reference the baseline sum LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions and no new lesions having appeared; SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum LD. PD defined as at least 20% increase in the sum of LD of target, lesions taking as reference, the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions or progression of nontarget lesions.
Time Frame: Randomization up to 37.52 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 118 | 118
percentage of participants | 71.2 [62.1 to 79.2] | 64.4 [55.1 to 73.0]

5. Secondary Outcome: Time to Progressive Disease (TtPD)
Description: TtPD was defined as the time from randomization to the first date of objectively determined progressive disease (PD). For participants who were not known to have had objective progression of disease as of the data-inclusion cut-off date for a particular analysis, or who had died without objective progression of disease, TtPD was censored at the date of the participant's last objective progression-free disease assessment prior to cut-off date.
Time Frame: Randomization to the first date of measured PD up to 37.32 months
Population: Intent-to-treat (ITT) population: All data from all randomized participants according to the treatment they were assigned. Censored participants: Pemetrexed + Cisplatin + Gefitinib (G) =37, G=26.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 118 | 118
months | 8.61 [6.60 to 11.20] | 9.69 [6.87 to 11.20]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin + Gefitinib vs Gefitinib; Test type: Superiority or Other; p = 0.252, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.63 to 1.14]

6. Secondary Outcome: Duration of Tumor Response
Description: The duration of a complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria was defined as the time from first objective status assessment of CR or PR to the first time of objective disease progression or death as a result of any cause. CR was defined as the disappearance of all tumor lesions. PR was defined as at least a 30% decrease in sum of longest diameter (LD) of target lesions taking as reference the baseline sum of LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions and no new lesions having appeared. Participants who were not known to have died or had objective progression of disease as of the data-inclusion cut-off date were censored at the date of the participant's last complete objective progression-free disease assessment prior to that cut-off date.
Time Frame: Date of initial response to the date of measured PD or death up to 34.43 months
Population: A subset of the Intent-to-treat (ITT) population: All data from all randomized participants according to the treatment they were assigned who had confirmed CR or PR. Pemetrexed + Cisplatin + Gefitinib= 19, Gefitinib= 9.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 49 | 56
months | 12.09 [7.16 to 22.11] | 11.93 [9.63 to 14.09]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin + Gefitinib vs Gefitinib; Test type: Superiority or Other; p = 0.952, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.53 to 1.32]

7. Secondary Outcome: Time to Worsening of Health-Related Quality of Life (TWQ) Using the Participant-Rated Lung Cancer Symptom Scale (LCSS)
Description: The LCSS data included participant ratings of 6 symptoms (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain) and 3 summary items (overall symptom severity, interference with daily activities, and overall QoL). Participants recorded their ratings for each item, by placing a mark on a visual analog scale (VAS) that ranged from 0 millimeter (mm) (lower symptom burden, less interference with normal activity, or better QoL) to 100 mm (higher symptom burden, more interference with normal activity, or worse QoL). TWQ was evaluated from date of randomization to first date of worsening, defined as a half standard deviation change as determined from the corresponding baseline item score in the pooled treatment group. For participants not known to have worsened or who were lost to follow-up, TWQ was censored at date of the participant's last LCSS assessment.
Time Frame: Every cycle while on-study therapy and at 3 months post last dose
Population: Participants who received at least 1 dose of study treatment and had LCSS data available. Participants censored (Pemetrexed + Cisplatin + Gefitinib, Gefitinib): Loss of appetite (33,59), Fatigue (42,54), Cough (52,65), Dyspnea (51,66), Hemoptysis (69,74), Pain (48,67), Overall symptoms (52,63), Interference (42,59), Overall QoL (51,51).
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Number analyzed (Participants) | 109 | 109
months
  Loss of appetite | 2.99 [1.71 to 3.68] | 7.95 [4.90 to NA] — upper bound not generated due to small sample size
  Fatigue | 4.83 [2.92 to 6.83] | 7.29 [3.75 to 13.63]
  Cough | 8.57 [5.68 to 10.94] | 16.69 [6.51 to NA] — upper bound not generated due to small sample size
  Dyspnea | 6.97 [3.15 to 15.44] | 18.23 [7.06 to NA] — upper bound not generated due to small sample size
  Hemoptysis | 19.45 [9.89 to NA] — upper bound not generated due to small sample size | 17.05 [10.02 to NA] — upper bound not generated due to small sample size
  Pain | 6.44 [2.92 to 11.40] | 15.57 [9.95 to NA] — upper bound not generated due to small sample size
  Overall symptoms | 4.76 [3.12 to 12.81] | 13.63 [7.06 to NA] — upper bound not generated due to small sample size
  Interference | 4.50 [3.02 to 7.03] | 8.34 [4.90 to NA] — upper bound not generated due to small sample size
  Overall quality of life | 6.14 [3.52 to 12.78] | 6.93 [3.22 to 13.63]

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to progressive disease were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Arm/Group | Pemetrexed + Cisplatin + Gefitinib | Gefitinib
Serious Adverse Events (participants affected / at risk) | 35/114 | 32/118
Other Adverse Events (participants affected / at risk) | 111/114 | 110/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pemetrexed + Cisplatin + Gefitinib (N=114) | Gefitinib (N=118)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 9 (9)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/84 (0) | 1/89 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin + Gefitinib (N=114) | Gefitinib (N=118)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 21 (46) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 13 (16) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 7 (11) | 2 (2)
Constipation (Gastrointestinal disorders) | 36 (52) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 30 (38) | 50 (68)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 70 (133) | 26 (27)
Stomatitis (Gastrointestinal disorders) | 10 (10) | 12 (16)
Vomiting (Gastrointestinal disorders) | 41 (69) | 13 (14)
Asthenia (General disorders) | 10 (10) | 3 (3)
Chest pain (General disorders) | 9 (10) | 7 (8)
Fatigue (General disorders) | 32 (49) | 21 (22)
Influenza like illness (General disorders) | 8 (18) | 6 (7)
Mucosal inflammation (General disorders) | 6 (8) | 12 (13)
Pyrexia (General disorders) | 8 (9) | 13 (16)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (7)
Paronychia (Infections and infestations) | 9 (14) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 8 (10)
Alanine aminotransferase increased (Investigations) | 20 (23) | 30 (33)
Aspartate aminotransferase increased (Investigations) | 16 (18) | 24 (30)
Blood creatinine increased (Investigations) | 6 (10) | 2 (3)
Haemoglobin decreased (Investigations) | 13 (15) | 4 (9)
Neutrophil count decreased (Investigations) | 14 (28) | 0 (0)
White blood cell count decreased (Investigations) | 8 (16) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 43 (57) | 29 (32)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 11 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 10 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (11) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Dizziness (Nervous system disorders) | 21 (22) | 16 (19)
Headache (Nervous system disorders) | 18 (23) | 16 (19)
Neuropathy peripheral (Nervous system disorders) | 14 (14) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (14) | 4 (5)
Insomnia (Psychiatric disorders) | 14 (14) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (33) | 21 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 20 (21)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 8 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 17 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (9)
Acne (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (18) | 9 (9)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 11 (12) | 20 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (12) | 25 (27)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (43) | 38 (47)
Rash (Skin and subcutaneous tissue disorders) | 36 (51) | 52 (72)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Hypertension (Vascular disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days